CLINICAL TRIAL: NCT00060554
Title: A Safety and Efficacy Trial Evaluating the Use of Fondaparinux in Percutaneous Coronary Intervention (PCI)(63133)(WITHDRAWN)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug sold to Sanofi-Aventis who sold it to GSK; OBS no longer owns study and does not have data.
Sponsor: Schering-Plough (Industry)
Responsible Party: Head, Clinical Trials Registry & Results Disclosure Group, Schering-Plough
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 63133 (ASPIRE-Pilot)
Record Dates: First submitted 2003-05-07; First posted 2003-05-08 (Estimated); Last update posted 2009-11-03 (Estimated); Status verified 2009-11

CONDITIONS: Myocardial Infarction; Coronary Disease
Keywords: Elective PCI; Heart catherization; Acute coronary syndromes
MeSH Terms: conditions — Myocardial Infarction; Coronary Disease; Acute Coronary Syndrome | interventions — Fondaparinux; Heparin; Percutaneous Coronary Intervention

INTERVENTIONS:
Drug: fondaparinux sodium
Drug: heparin
Procedure: percutaneous coronary intervention (PCI)

SUMMARY:
The purpose of this research study is to obtain experience in the use of fondaparinux (Arixtra) as compared to heparin when administered to patients who undergo percutaneous coronary intervention (PCI). PCI is a mechanical procedure used to widen the narrowing in a coronary artery in patients with symptomatic coronary artery disease. Fondaparinux and heparin are drugs that inhibit blood clotting.

ELIGIBILITY:
Inclusion criteria

* Scheduled for PCI, including PCI for non-ST elevation acute coronary syndromes (ACS), primary PCI for ST elevation myocardial infarction (MI) or elective PCI (with planned overnight stay in hospital). (Patients undergoing diagnostic heart catherization who are suitable candidates for "ad hoc" PCI are also eligible).

Exclusion criteria:

* Age < 21 years
* Activated Clotting Time (ACT) > 200 seconds immediately prior to PCI
* Use of low molecular weight heparin (LMWH) in the previous 6 hours before PCI
* Currently receiving an oral anticoagulant (OAC) agent with an INR > 1.8
* Thrombolytic therapy for ST elevation MI in the previous 24 hours before PCI
* Active internal bleeding or history of hemorrhagic diathesis
* Thrombocytopenia (platelet count < 100 x 10-9/L)
* Pregnant women or women of childbearing potential who are not using an effective method of contraception
* Known allergy to unfractionated heparin, fondaparinux, aspirin or clopidogrel
* Absolute contra-indication to anticoagulation
* Participation in other clinical research studies involving the evaluation of other investigational drugs or devices within 30 days of enrollment or prior participation in this study.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300
Dates: Start 2003-04

CONTACTS AND LOCATIONS:
Locations (26):
- United States (8):
  - Ocala Research Institute, Inc., Ocala, Florida
  - University of Chicago - Section of Cardiology, Chicago, Illinois
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan, Dept. of Internal Medicine, Ann Arbor, Michigan
  - Greenville Hospital System, Greenville, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - The Methodist Hospital, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- Canada (11):
  - Foothills Hospital, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Hospital & Health Sciences Centre, Vancouver, British Columbia
  - QE II Health Sciences Centre, New Halifax Infirmary, Halifax, Nova Scotia
  - HGH-McMaster Clinic, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Sunnybrook & Women's College Health Sciences Center, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Hopital du Sacre-Coeur de Montreal, Montreal, Quebec
- France (7):
  - Hopital Jean Minjoz, Besançon, Cedex
  - CHU de Caen, Caen, Cedex
  - Hopital du Bocage, Dijon, Cedex
  - CHU de Rangueil, Toulouse, Cedex
  - Centre Hospitalier de Lagny-Marne La Vallee, Lagny, Sur Marne
  - Hopital Europeen Georges Pompidou, Paris
  - Hopital Bichat, Paris